CLINICAL TRIAL: NCT07244367
Title: Maintenance Venetoclax Based Therapy Post Complete Remission in AML Fit Patients
Brief Title: Maintenance Venetoclax in AML Fit Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Ibrahim Abdelshakour, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-25-9---3MD
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukaemia (AML)
Keywords: AML; Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: this study is a prospective,phase III , randomized ,open , interventional study. double blind, placebo control clinical trial . Evaluating efficacy of maintenance venetoclax based therapy in Acute meyloid leukemia fit patients who acheived complete remission after standard induction and consolidation therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): will receive SC cytarabine + venetoclax till bone marrow transplantation or for 12 cycles for patient will not undergo BMT , SC Cytarabine (20 mg) administrated on days 1-7 , Venetoclax (100 mg ) administrated on days 1-7 , Voriconazole 200 mg 1x2 administrated on days 1-7 + best supportive care BSC
  Interventions: Drug: SC cytarabine +Venetoclax
- Arm B (No Intervention): Patients Will receive Best supportive care( BSC )only

INTERVENTIONS:
Drug: SC cytarabine +Venetoclax — SC Cytarabine (20 mg) administrated on days 1-7 ,,Venetoclax (100 mg ) administrated on days 1-7,,Voriconazole 200 mg 1x2 administrated on days , Best supportive care as needed . Up to 12 cycles or until patients undergo bone marrow transplantation
  Other Names: Venclexta
  Arms: Arm A

SUMMARY:
this study will explore the efficacy of maintenance SC cytarabine + venetoclax therapy as regard disease free survival (DFS) in AML fit patients who achieved CR after highly aggressive chemotherapy as bridge for BMT or if BMT will be delayed or canceled due to any other reason.

DETAILED DESCRIPTION:
this study is a prospective,phase III , randomized ,open , interventional study include young fit patients who will receive maintenance venetoclax +subcutaneous cytarabine as bridge for BMT or if BMT will be delayed

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 - 60 years . Patients who are not eligible for immediate bone marrow transplantation. Newly diagnosed AML patients who attained CR after 1st line. Refractory / recurrant AML patients who attained CR after 2nd line .

Exclusion Criteria:

* Patients not on CR . Age : younger than 18 or older than 60 . Patients not eligible for bone marrow transplation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival DFS | 24 months
  time from complet remission to relapse or death from any cause in AML fit patients receiving maintenance SC cytarabine plus venetoclax after intensive chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed M Ali, Professor, Study Director — Faculty of medicine sohag university
Locations (2):
- Egypt (2):
  - Sohag university hospital, Sohag
  - Sohag university, Sohag

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Papaemmanuil E, Gerstung M, Bullinger L, Gaidzik VI, Paschka P, Roberts ND, et al. Genomic classification and prognosis in acute myeloid leukemia. N Engl J Med. 2016;374:2209-21. 2. DiNardo CD, Erba HP, Freeman SD, Wei AH. Acute myeloid leukaemia. Lancet. 2023;401:2073-86. 3. Miranda-Filho A, Piñeros M, Ferlay J, et al: Epidemiological patterns of leukaemia in 184 countries: A population-based study. Lancet Haematol 5:e14-e24, 2018